CLINICAL TRIAL: NCT00800904
Title: Asthma Control Among Patients Who Were Receiving Inhaled Corticosteroids in General Practice in Thailand
Brief Title: Asthma Control Among Patients Receiving Inhaled Corticosteroids in Thailand
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Thanu Komolsai, MD, Medical Advisor, AstraZeneca (Thailand) Ltd.
Other Study IDs: NIS-RTH-DUM-2008/1
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Asthma
Keywords: Asthma; Inhaled corticosteroid; Thai patient eligibility; Persistent asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the percentage of patients who has reached the GINA guideline of asthma treatment after receiving any inhaled corticosteroid for 3 months or longer in actual clinical practice. Such percentage for each level of severity - mild, moderate and severe persistent asthma as well as the differences of these rates will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Established persistent asthma
* Currently treated with any inhaled corticosteroid therapy but not SYMBICORT nor SERETIDE for 3 months or longer

Exclusion Criteria:

* Currently participating or have participated in a study with an investigational compound within the last 30 days
* Current diagnosis of chronic obstructive pulmonary disease (COPD)
* Smoked more than 10 packs a year

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient aged 12 years and older who established persistent asthma and currently treated with any inhaled corticosteroid for 3 months or longer.
Sampling Method: Non-Probability Sample
Enrollment: 1210 (Estimated)
Dates: Start 2009-05; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Asthma control test | On the survey date

SECONDARY OUTCOMES:
Asthma control in mild, moderate and severe persistent asthma patients | On the survey date

CONTACTS AND LOCATIONS:
Overall Officials: Bandit Thinkhamrop, PhD, Principal Investigator — Department of Biostatistics and Demography, Faculty of Public Health, Khon Kaen University; Watchara Boonsawat, MD. PhD, Principal Investigator — Department of Medicine, Faculty of Medicine, Khon Kaen University
Locations (26):
- Thailand (26):
  - Research Site, Amnat Charoen
  - Research Site, Buriram
  - Research Site, Chachoengsao
  - Research Site, Chaiyaphum
  - Research Site, Chanthaburi
  - Research Site, Chiang Rai
  - Research Site, Kalasin
  - Research Site, Khon Kaen
  - Research Site, Lopburi
  - Research Site, Mae Hong Son
  - Research Site, Mahasarakham
  - Research Site, Nakhon Phanom
  - Research Site, Nakhorn Ratchasima
  - Research Site, Nan
  - Research Site, Nong Khai
  - Research Site, Samutsongkhram
  - Research Site, Si Sa Ket
  - Research Site, Sing Buri
  - Research Site, Songkhla
  - Research Site, Sukhothai Thani
  - Research Site, Surat Thani
  - Research Site, Trang
  - Research Site, Trat
  - Research Site, Ubon Ratchathani
  - Research Site, Udon Thani
  - Research Site, Yasothon